CLINICAL TRIAL: NCT00763802
Title: Validation of a Predictive Model to Estimate the Risk of Conversion to Clinically Significant Macular Edema and/or Vision Loss in Mild Nonproliferative Diabetic Retinopathy in Diabetes Type 2
Acronym: CPM
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Other Study IDs: PTDC/SAU-OSM/72635/2006
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- MNPDR: Type 2 diabetic patients with Mild non-prolipherative retinopathy.

SUMMARY:
This project aims to validate a predictive model of diabetic retinopathy progression to clinically significant macular edema (CSME) needing photocoagulation and/or vision loss. The Coimbra Predictive Model (CPM), based on retinal thickness, microaneurysms number, HbA1C and LDL levels, established on a set of 52 diabetic patients, will be tested on a population of 400 patients/eyes to be enrolled into the study. These patients will perform 2 visits at 6-month interval (V0 and V6) to classify each patient into one of the 3 previously established phenotypes. Two years after (V24) patients will be reexamined. The occurrence of end-points, achieved by the patients, are expected to validate our predictive model.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2 according to 1985 WHO criteria.
* Age between 35 and 75 years.
* Mild non-prolipherative retinopathy (based on ETDRS criteria)
* Best Corrected Visual acuity >20 /25
* Refraction with a spherical equivalent less than 5 Dp.
* Inform consent

Exclusion Criteria:

* Cataract or other eye disease that may interfere with fundus examinations
* Glaucoma
* Vitreous syneresis or posterior vitreous detachment
* Other retinal vascular disease
* Recent intraocular surgery
* Previous laser therapy
* Dilatation of the pupil < 5 mm

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients with Mild non-prolipherative retinopathy fulfilling the inclusion criterion.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
CSME needing Photocoagulation | 24 months

SECONDARY OUTCOMES:
Vision Loss | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: José G Cunha-Vaz, MD, PhD, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI, Coimbra, Coimbra District, Portugal

REFERENCES:
- [Background] Cunha-Vaz J, Bernardes R. Nonproliferative retinopathy in diabetes type 2. Initial stages and characterization of phenotypes. Prog Retin Eye Res. 2005 May;24(3):355-77. doi: 10.1016/j.preteyeres.2004.07.004. Epub 2004 Dec 16. PMID 15708833
- [Background] Lobo CL, Bernardes RC, Figueira JP, de Abreu JR, Cunha-Vaz JG. Three-year follow-up study of blood-retinal barrier and retinal thickness alterations in patients with type 2 diabetes mellitus and mild nonproliferative diabetic retinopathy. Arch Ophthalmol. 2004 Feb;122(2):211-7. doi: 10.1001/archopht.122.2.211. PMID 14769598
- [Background] Hayreh SS. Diabetic papillopathy and nonarteritic anterior ischemic optic neuropathy. Surv Ophthalmol. 2002 Nov-Dec;47(6):600-2; author reply 602. doi: 10.1016/s0039-6257(02)00358-2. No abstract available. PMID 12504747
- [Background] Pires I, Bernardes RC, Lobo CL, Soares MA, Cunha-Vaz JG. Retinal thickness in eyes with mild nonproliferative retinopathy in patients with type 2 diabetes mellitus: comparison of measurements obtained by retinal thickness analysis and optical coherence tomography. Arch Ophthalmol. 2002 Oct;120(10):1301-6. doi: 10.1001/archopht.120.10.1301. PMID 12365908
- [Derived] Cunha-Vaz J, Ribeiro L, Costa M, Simo R. Diabetic Retinopathy Phenotypes of Progression to Macular Edema: Pooled Analysis From Independent Longitudinal Studies of up to 2 Years' Duration. Invest Ophthalmol Vis Sci. 2017 May 1;58(6):BIO206-BIO210. doi: 10.1167/iovs.17-21780. PMID 28785768
- [Derived] Cunha-Vaz J, Ribeiro L, Lobo C. Phenotypes and biomarkers of diabetic retinopathy. Prog Retin Eye Res. 2014 Jul;41:90-111. doi: 10.1016/j.preteyeres.2014.03.003. Epub 2014 Mar 26. PMID 24680929
- [Derived] Pires I, Santos AR, Nunes S, Lobo C, Cunha-Vaz J. Subclinical macular edema as a predictor of progression to clinically significant macular edema in type 2 diabetes. Ophthalmologica. 2013;230(4):201-6. doi: 10.1159/000354550. Epub 2013 Sep 25. PMID 24080704
- [Derived] Nunes S, Ribeiro L, Lobo C, Cunha-Vaz J. Three different phenotypes of mild nonproliferative diabetic retinopathy with different risks for development of clinically significant macular edema. Invest Ophthalmol Vis Sci. 2013 Jul 10;54(7):4595-604. doi: 10.1167/iovs.13-11895. PMID 23745006
- [Derived] Pires I, Santos AR, Nunes S, Lobo C. Macular thickness measured by stratus optical coherence tomography in patients with diabetes type 2 and mild nonproliferative retinopathy without clinical evidence of macular edema. Ophthalmologica. 2013;229(4):181-6. doi: 10.1159/000350593. Epub 2013 Apr 24. PMID 23614970
- [Derived] Ribeiro ML, Nunes SG, Cunha-Vaz JG. Microaneurysm turnover at the macula predicts risk of development of clinically significant macular edema in persons with mild nonproliferative diabetic retinopathy. Diabetes Care. 2013 May;36(5):1254-9. doi: 10.2337/dc12-1491. Epub 2012 Nov 30. PMID 23204247
- See also: Related Info — http://www.aibili.pt